CLINICAL TRIAL: NCT03791996
Title: Impact of Cranioplasty on Cognitive Outcome: A Multi-Center Prospective Randomized Study
Brief Title: Cranioplasty Cognitive Outcome Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kwong Wah Hospital (Other)
Collaborators: The Queen Elizabeth Hospital (Other); Queen Mary Hospital, Hong Kong (Other); Prince of Wales Hospital, Shatin, Hong Kong (Other); Princess Margaret Hospital, Canada (Other); Tuen Mun Hospital (Other Government); Pamela Youde Nethersole Eastern Hospital (Other)
Responsible Party: Principal Investigator, Peter Woo Yat Ming, Principal Investigator, Kwong Wah Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCO-RCT
Record Dates: First submitted 2018-12-30; First posted 2019-01-03 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Cognitive Impairment; Brain Herniation
Keywords: Cranioplasty; Craniectomy; Cognitive impairment; Syndrome of the trephined
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: 2-arm randomised study with subjects centrally randomised by assigning them into either the control "late" cranioplasty group or the intervention "early" cranioplasty group.
  All subjects will eventually receive the cranioplasty procedure.
Masking Description: 1:1 block central randomisation with assignments written on a card sealed in an opaque envelop.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Late" cranioplasty (No Intervention): Subjects undergoing cranioplasty within 3 months after craniectomy.
- "Early" cranioplasty (Experimental): Subjects undergoing cranioplasty beyond 3 months after craniectomy.
  Interventions: Procedure: "Early" cranioplasty

INTERVENTIONS:
Procedure: "Early" cranioplasty — Subjects undergoing cranioplasty beyond 3 months after craniectomy.
  Arms: "Early" cranioplasty

SUMMARY:
This will be a multicenter prospective randomized study of adult patients with an acquired skull defect as a result of craniectomy and considered suitable for cranioplasty, i.e. reconstruction of the skull defect, at all seven Hong Kong Hospital Authority neurosurgical units. Patients that underwent their primary craniectomy operation at any of the Hospital Authority neurosurgery centers from the 1st March 2019 and considered suitable for cranioplasty will be included in this study. Those who underwent their primary craniectomy before 1st March 2019 or at an institution other than the aforementioned neurosurgical units will be excluded. Data from clinical records, operation notes, medication-dispensing records, laboratory records and radiological reports will be collected.

30 adult patients with craniectomy will be recruited and randomized into two groups: "early" cranioplasty, i.e. performed within 3 months of craniectomy, and "late", i.e. cranioplasty performed more than 3 months after the operation. The aim of the study is to determine whether early cranioplasty can improve on patient's cognitive performance compared to those who undergo the procedure after 3 months.

DETAILED DESCRIPTION:
Decompressive craniectomy, a neurosurgical procedure where a portion of the skull calvarium is removed, is a life-saving procedure. The complication rate of cranioplasty, a neurosurgical procedure where the acquired skull defect is reconstructed, ranges from 11% to 26% and includes postoperative hemorrhage and infection. (4) The syndrome of the trephined is a recognized long-term complication in which certain groups of patients, experience debilitating neurocognitive deficits in addition to chronic headache, dizziness, fatigability and clinical depression. (2) It is believed that the lack of an overlying bone may cause undue significant atmospheric pressure on the underlying cortex, thereby reducing cerebral perfusion and cerebrospinal fluid flow. There are reports that cognitive improvement can be observed in up to 30% of patients after cranioplasty yet the underlying mechanism for this observation is unclear. (1) Some studies have demonstrated enhanced cerebral perfusion by non-invasive investigations, but there is a lack of large scale systematically performed studies to verify such cerebral hemodynamic effects. (1-3) Clinical equipoise exists regarding the optimum timing of cranioplasty procedures after craniectomies. While the anecdotal practice of delaying cranioplasty for at least 3 months after a craniectomy is common, local and overseas observational studies suggest that performing early cranioplasties (i.e. within 3 months) is equally safe in terms of infection and other operative complications. (4-6)

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years-old,
2. Craniectomy was performed due to head injury, infarct or spontaneous intracerebral hemorrhage, and benign tumors.
3. Craniectomy skull defect size of >10cm at its longest diameter
4. Craniectomy performed at any of the Hospital Authority's Neurosurgical Centers after 1st March 2019

Exclusion Criteria:

1. Age older than 80 years-old,
2. Patients cannot communicate by obeying simple command,
3. Patients who are unfit for cranioplasty as decided by the treating neurosurgeon
4. Posterior fossa craniectomy
5. Craniectomy performed before 1st March 2019
6. Craniectomy performed at an institution outside the Hospital Authority
7. Any pre-existing illness that renders the patient moderately or severely disabled before the brain insult.
8. Patients that need an additional procedure e.g. cerebrospinal fluid shunting with cranioplasty in the same setting.
9. History of central nervous system infection
10. Craniectomy-related complications such as hemorrhage or surgical site infection requiring surgical intervention or deemed to affect patient's long-term cognitive outcome
11. Claustrophobia or any other medical condition that prohibits the patient from undergo MRI scanning
12. Patients who cannot understand spoken English or Chinese

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MOCA) | 3-months
  Minimum (worse): 0/30; Maximum (best) 30/30. Higher values represent a better outcome.
Neurobehavioural Cognitive State Examination (NCSE) | 3-months
  Multi-domain assessment involving: orientation, attention, registration, comprehension, repetition, naming, construction, calculation, similarities,judgement. Stratification of each domain into mild, moderate and severe impairment. The higher the number the better the outcome.
Rivermead Behavioural Memory Test (RBMT) | 3-months

SECONDARY OUTCOMES:
Motor assessment | 3-months
  Medical Research Council limb power
Modified Functional Ambulation Category (MFAC) | 3-months
  7 ordinal scale assessment. The lower the scale, the worse the ambulatory ability of the patient. I: bed bound; 2: wheel-chair bound; 3: dependent walker; 4: Assisted walker; 5: Supervised walker; 6: Indoor walker; 7: Outdoor walker (patient can walk anywhere).
Quality of life assessment | 3-months
  Short Form-36 (SF-36)
Psychological assessment | 3-months
  Beck depression inventory (BDI)
Caregiver assessment | 3-months
  Caregiver Strain Index
Caregiver | 3-months
  Caregiver self-assessment questionnaire
MRI cerebral perfusion assessment | 3-months
  Cerebral blood flow

CONTACTS AND LOCATIONS:
Overall Officials: Calvin Mak, MBBS FRCS, Principal Investigator — Neurosurgery, Queen Elizabeth Hospital
Locations (1):
- Kwong Wah Hospital, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Halani SH, Chu JK, Malcolm JG, Rindler RS, Allen JW, Grossberg JA, Pradilla G, Ahmad FU. Effects of Cranioplasty on Cerebral Blood Flow Following Decompressive Craniectomy: A Systematic Review of the Literature. Neurosurgery. 2017 Aug 1;81(2):204-216. doi: 10.1093/neuros/nyx054. PMID 28368505
- [Result] Bender A, Heulin S, Rohrer S, Mehrkens JH, Heidecke V, Straube A, Pfefferkorn T. Early cranioplasty may improve outcome in neurological patients with decompressive craniectomy. Brain Inj. 2013;27(9):1073-9. doi: 10.3109/02699052.2013.794972. Epub 2013 May 10. PMID 23662672
- [Result] Ashayeri K, M Jackson E, Huang J, Brem H, Gordon CR. Syndrome of the Trephined: A Systematic Review. Neurosurgery. 2016 Oct;79(4):525-34. doi: 10.1227/NEU.0000000000001366. PMID 27489166
- [Result] Malcolm JG, Rindler RS, Chu JK, Grossberg JA, Pradilla G, Ahmad FU. Complications following cranioplasty and relationship to timing: A systematic review and meta-analysis. J Clin Neurosci. 2016 Nov;33:39-51. doi: 10.1016/j.jocn.2016.04.017. Epub 2016 Aug 4. PMID 27499122
- [Result] Xu H, Niu C, Fu X, Ding W, Ling S, Jiang X, Ji Y. Early cranioplasty vs. late cranioplasty for the treatment of cranial defect: A systematic review. Clin Neurol Neurosurg. 2015 Sep;136:33-40. doi: 10.1016/j.clineuro.2015.05.031. Epub 2015 May 29. PMID 26056810
- [Result] Tsang AC, Hui VK, Lui WM, Leung GK. Complications of post-craniectomy cranioplasty: risk factor analysis and implications for treatment planning. J Clin Neurosci. 2015 May;22(5):834-7. doi: 10.1016/j.jocn.2014.11.021. Epub 2015 Mar 28. PMID 25827865